CLINICAL TRIAL: NCT06035679
Title: Prospective, Single-center, Observational Clinical Study of Pyrotinib Combined With Trastuzumab and Chemotherapy Neoadjuvant Therapy for HER2-positive Breast Cancer
Brief Title: Pyrotinib Combined With Trastuzumab and Chemotherapy Neoadjuvant Therapy for HER2-positive Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Youzhi Zhu (Other)
Responsible Party: Sponsor-Investigator, Youzhi Zhu, Clinical Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-95
Record Dates: First submitted 2023-08-31; First posted 2023-09-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib Combined With Trastuzumab and Chemotherapy (Experimental): T1cN0M0 HER2+ breast cancer Patients received 2 cycles (pyrotinib + trastuzumab + taxoid) regimen and were evaluated to continue with the original regimen if PR, and 4 cycles (pyrotinib + trastuzumab + taxoid + carboplatin) regimen if SD/PD. Phase II-III HER2+ breast cancer Patients received 6 cycles of treatment (pyrotinib + trastuzumab + taxoid + carboplatin)
  Interventions: Drug: Pyrotinib and Trastuzumab

INTERVENTIONS:
Drug: Pyrotinib and Trastuzumab — Small and large molecules combined with chemotherapy for neoadjuvant treatment of HER2-positive breast cancer
  Other Names: dual HER2 blockade in the neoadjuvant setting

SUMMARY:
This study is a prospective, single-center, observational clinical study, The objection was to observe the treatment of pyrotinib combined with trastuzumab and neoadjuvant chemotherapy Efficacy of Stage II-III breast cancer and observation of the efficacy of step-down neoadjuvant therapy for HER2-positive stage T1cN0M0 breast cancer.

DETAILED DESCRIPTION:
This study is a prospective, single-center, observational clinical study,Which plan to be enroll 30 patients with HER2-positive early breast cancer receive pyrotinib combined with trastuzumab and chemotherapy neoadjuvant therapy. The primary endpoint was the total pathological complete response rate (tpCR) , The objection was to observe the treatment of pyrotinib combined with trastuzumab and neoadjuvant chemotherapy Efficacy of Stage II-III breast cancer and observation of the efficacy of step-down neoadjuvant therapy for HER2-positive stage T1cN0M0 breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years;
2. Her2-positive breast cancer confirmed by pathology;
3. invasive breast cancer confirmed by histology, Tumor stage: early stage (T1c-3, N0-1, M0) or locally advanced stage (T2-4, N2, N3, M0);
4. ECOG PS: 0-1 score;
5. Plan to undergo the final surgical removal of breast cancer, i.e. breast conserving surgery or total mastectomy, sentinel lymph node (SN) biopsy or axillary lymph node dissection (ALND)
6. Normal function of major organs means that the following criteria are met:

(1) Blood test neutrophil (ANC) >=1.5x10^9/L; Platelet count (PLT) >=90x10^9/L; Hemoglobin (Hb) >=90g/L; (2) Total bilirubin (TBIL) <=1.5 upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=1.5xULN; Alkaline phosphatase <=2.5xULN; Urea nitrogen (BUN) and creatinine (Cr) <=1.5xULN; (3) Left ventricular ejection fraction (LVEF) >=55%; (4) The QT interval (QTcF) corrected by Fridericia method was less than 470msec in 12-lead ECG; 7. For women who have not undergone menopause or surgical sterilization: consent to abstinence or use an effective contraceptive method (during treatment and for at least 7 months after the last dose in the study treatment); 8. Volunteer to participate in this study, sign the informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Known allergic history of the drug components of this protocol;
2. Previous or co-existing other malignant tumors, except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
3. Participated in clinical trials of other antitumor drugs within four weeks;
4. Stage IV (metastatic) breast cancer;
5. Multiple factors affecting oral medication (e.g., inability to swallow, post-gastrointestinal resection, chronic diarrhea, and intestinal obstruction);
6. A history of congestive heart failure (CHF) or uncontrolled heart disease (angina, arrhythmia, hypertension);
7. Patients with active infection and severe mental illness;
8. Pregnant or lactating patients;
9. Patients with allergies or known history of allergies to the drug components of this protocol; A history of immunodeficiency, including being HIV positive, or having other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
10. Concomitant diseases that, in the judgment of the investigator, seriously endanger the patient's safety or interfere with the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
tpCR | at surgery
  total Pathological Complete Response

CONTACTS AND LOCATIONS:
Overall Officials: zhu youzhi, Study Chair — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujan Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available